CLINICAL TRIAL: NCT05205694
Title: Biomarkers of Oral Health in Covid-19 Survivors
Brief Title: Oral Health in Covid-19 Survivors
Acronym: ORFCovid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Jelena Roganović, Associate Professor, University of Belgrade
Other Study IDs: 36/10
Record Dates: First submitted 2022-01-22; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-09

CONDITIONS: COVID-19; Periodontitis
MeSH Terms: conditions — COVID-19; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Late COVID-19 and PERIO: Participants in the late convalescent stage of COVID-19 with diagnosed periodontitis
- PERIO non COVID-19: Participants with diagnosed periodontitis and no history of COVID-19
- Late COVID-19 non PERIO: Participants in the late convalescent stage of COVID-19 without periodontitis
- Non PERIO non COVID-19: Participants with no history of COVID-19 and without periodontitis

SUMMARY:
Aims are to assess periodontal health and salivary stress/ immunity responses in COVID-19 survivors

DETAILED DESCRIPTION:
There are lack of data concerning oral health in COVID-19 survivors, nevertheless, many middle-aged patients with oral symptoms of Post-acute COVID-19 report xerostomia and taste impairment and suffer from oral hypofunction, thus may be susceptible to periodontitis and oral frailty. Post-acute or long COVID-19 is/would be the health hallmark of post-COVID-19 era, manifested as a multiplicity of clinical problems and requiring conceptual framework aiming at multidisciplinary health preserving activities. There are various factors which may affect oral and periodontal health in post-COVID-19 era, such as disruption of dental professional care due to the fear of infection, virus-induced disturbance of oral homeostasis and, as a common denominator- COVID-19-induced psychological stress. Expected results would not just offer epidemiological data but also, mechanistic background for defining risks and modified measures aiming to preserve oral health in post-COVID-19 era.

ELIGIBILITY:
Inclusion Criteria:

* self-reported good general health, ≥ 14 erupted teeth excluding third molars. For periodontally healthy: Bleeding on probing score ≤10%, without attachment loss and radiographic bone loss and probing depth ≤ 3 mm in every site (Trombelli L et al., 2018). For periodontitis patients: periodontitis in stages II-IV.

Exclusion Criteria:

* history of periodontal treatment in previous six months, acute oral infection, presence of systemic disease(s), pregnancy, lactation, smoking ≥ 10 cigarettes per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Groups I and III will include COVID-19 survivors in late convalescent stage (one to six months post onset of symptoms accompanied by SARS-CoV-2- positive nasopharyngeal swab result) who had non-severe COVID-19 (no or mild pneumonia - less than 50 percent lung involvement on imaging within 24 to 48 hours, absence of dyspnea and hypoxia). Groups II and IV will include participants who report to had no symptoms of COVID-19 and had no SARS-CoV-2- positive nasopharyngeal swab result
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Periodontal disease stage and COVID 19 | one to six months after COVID-19
  Correlation periodontitis and COVID 19 infection

SECONDARY OUTCOMES:
Oral frailty | one to six months after COVID-19
  Oral frailty assessment in Covid 19 and Perio affected patients
psychological stress | one to six months after COVID-19
  Assessment of psychological stress
salivary stress/immunity mediators | one to six months after COVID-19
  Association of salivary stress/immunity mediators levels with perio disease in COVID 19 patients

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine University of Belgrade, Belgrade, Serbia